CLINICAL TRIAL: NCT00020735
Title: A Phase II Randomized Controlled Clinical Trial Of The Antiestrogen GTx-006 In Subjects With Prostate Cancer
Brief Title: Toremifene Followed by Radical Prostatectomy in Treating Patients With Stage I or Stage II Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joel Nelson, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Joel Nelson, MD, Professor and Chairman, Department of Urology, University of Pittsburgh School of Medicine; Chief, Division of Surgery, UPMC Shadyside Hospital, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PCI-00-105; CDR0000068708 (Registry Identifier: PDQ (Physician Data Query)); PCI-N01-CN-75018; NCI-P01-0181
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Toremifene; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral toremifene (Experimental)
  Interventions: Drug: toremifene; Procedure: neoadjuvant therapy
- observation (Other)
  Interventions: Procedure: conventional surgery

INTERVENTIONS:
Drug: toremifene
  Arms: oral toremifene
Procedure: conventional surgery
  Arms: observation
Procedure: neoadjuvant therapy
  Arms: oral toremifene

SUMMARY:
RATIONALE: Androgens can stimulate the growth of prostate cancer cells. Hormone therapy using toremifene may fight prostate cancer by reducing the production of androgens.

PURPOSE: Randomized phase II trial to study the effectiveness of toremifene followed by radical prostatectomy in treating patients who have stage I or stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the percent of high-grade prostatic intraepithelial neoplasia (HGPIN) present in the radical prostatectomy tissue (excluding the luminal area) of patients with stage I or II adenocarcinoma of the prostate treated with toremifene vs observation alone followed by radical prostatectomy.
* Compare the absolute and relative changes in HGPIN in patients treated with toremifene vs observation alone.
* Compare biomarkers (including DNA ploidy and nuclear morphology; Ki67 and MIB-1 expression; bcl-2 expression; frequency of cells expressing apoptotic bodies; microvessel density; and intraprostatic testosterone, dihydrotestosterone (DHT), and estradiol) in the radical prostatectomy tissue of patients treated with toremifene vs observation alone.
* Compare changes from baseline in serum biomarkers, particularly PSA and hormone profiles (testosterone, DHT, androstenedione, dehydroepiandrosterone, androstanediol-glucuronide, estradiol, and sex hormone binding globulin), in patients treated with toremifene vs observation alone.
* Compare the safety of toremifene in these patients.
* Determine the relationships among pairs of biomarkers, biomarker changes, and outcome measures, including toxicity of toremifene and posttreatment HGPIN in these patients.
* Determine the relationship between HGPIN or biomarker responses and antiandrogen germline CAG repeat length polymorphism in patients treated with toremifene.
* Compare the tumor volume, margin status, and pT stage in patients treated with toremifene vs observation alone.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to participating center and baseline high-grade prostatic intraepithelial neoplasia (none vs more than 0% up to 10% vs more than 10%). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral toremifene daily for 3-6 weeks in the absence of unacceptable toxicity.
* Arm II: Patients undergo observation alone. Patients in both arms then undergo radical prostatectomy.

PROJECTED ACCRUAL: A total of 78 patients (52 for arm I, 26 for arm II) will be accrued for this study at a rate of 6-7 patients per month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Organ-confined (cT1-2) disease (stage I or II)
  * Must be schedule to undergo radical prostatectomy
  * Prior sextant biopsy required

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* ALT and AST less than 2 times ULN
* Alkaline phosphatase less than 2 times ULN
* No chronic hepatitis or cirrhosis

Renal:

* Creatinine less than 1.5 times ULN

Other:

* No severe mental or physical illness that would preclude radical prostatectomy
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* At least 5 years since prior antiestrogen, antiandrogen, LHRH agonist, estrogen, or progestational agent

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2001-04; Primary Completion 2005-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Percent of radical prostatectomy tissue volume (exclusive of luminal area) with high-grade prostatic intraepithelial neoplasia (HGPIN) present

CONTACTS AND LOCATIONS:
Overall Officials: Joel B. Nelson, MD, Study Chair — University of Pittsburgh
Locations (1):
- Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States